CLINICAL TRIAL: NCT04786522
Title: Influence of Irisin on Muscle Quality in a Cohort of Charcot-Marie-Tooth Patients
Brief Title: Irisin Levels in Patients With Charcot-Marie-Tooth (CMT) Disease
Acronym: IRICDE
Status: Completed | Type: Observational
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Michele Barone, Professor, University of Bari
Other Study IDs: Iri-mCMT
Record Dates: First submitted 2021-03-01; First posted 2021-03-08 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Charcot-Marie-Tooth Disease
Keywords: bioimpedance analysis; handgrip strength; body composition
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bioimpedenziometry, Handgrip strenght evaluation — The measurement of body composition was performed using Bioimpedance (BIA 101, Akern srl, Pontassieve (FI), Italy). The handgrip dynamometer (Jamar, Sammons Preston, Bolingbrook, IL, USA) was used to determine the isometric force of the forearm.
Diagnostic Test: Evaluation on blood specimens — Serum samples were assayed for calcium, phosphorus, magnesium, iron, lactate dehydrogenase (Ldh), creatine phosphokinase (Cpk), creatine kinase myocardial band (Ckmmb), myoglobin, thyroid stimulating hormone (TSH), 25(OH)-Vitamin D, osteocalcin, bone alkaline phosphatase (b-ALP), C-terminal telopeptide of type I collagen (CTX-I), haptoglobin, sclerostin, myostatin, and Irisin. Irisin serum concentrations were detected using a competitive ELISA kit (AdipoGen, Liestal, Switzerland)

SUMMARY:
Irisin is an exercise-mimetic myokine secreted by skeletal muscle. Compelling evidence in animal models and humans showed that Irisin prevents onset of musculoskeletal atrophy and its low serum levels are predictive of sarcopenia. The investigators evaluated the levels of irisin in patients affected by an hereditary motor and sensory neuropathy, namely Charcot-Marie-Tooth disease (CMT), in order to investigate possible key determinants of their muscle quality and possibly prevent the progressive distal weakness and muscle atrophy.

DETAILED DESCRIPTION:
Currently, there are no effective treatment approaches for CMT other than treating symptoms with medications such as nonsteroidal anti-inflammatory drugs that provide relief of lower back or leg pain. Except for the most severe cases in which orthopedic surgery is recommended to correct pes cavus and/or spine deformities, rehabilitative management of patients with CMT has shown that physical activity can provide a moderate increase in muscle strength and musculoskeletal function, improving activities of daily living. Benefits of exercise on the musculoskeletal system are widely recognized as primary non-pharmacologic intervention for several diseases. The positive outcome of physical activity is achieved not only by the mechanical load applied on the musculoskeletal system, but also via biochemical signals, the myokines, secreted during contraction that act locally or systemically on several body districts. Among these, Irisin is a hormone-peptide synthesized from skeletal muscle performing key actions on the whole-body metabolism. In humans, the investigators have documented with several studies an existing positive association between circulating levels of Irisin and bone mineral density. Very recently, in muscle biopsies of older adult subjects, the investigators also observed that the expression of the Irisin precursor, the fibronectin type III domain-containing protein 5 (FNDC5), was positively associated with Irisin serum levels and osteocalcin mRNA expression in bone biopsies, indicating a strong correlation between healthy muscle and bone tissues. In humans, low levels of circulating Irisin have been found to be predictive of muscle weakness and atrophy, and Irisin has been identified as a sensitive molecular biomarker for sarcopenia in postmenopausal women. In addition, women older than 65 years undergoing a 12-week exercise program showed an increase in circulating Irisin and an improvement in isokinetic leg strength and grip strength compared with control women. Moreover, there was a positive correlation between Irisin levels with grip strength and leg strength in the exercise group, suggesting a causal relationship between improved muscle strength and increased Irisin concentration. Although numerous reports recommend increasing muscle strength in CMT patients to prevent progressive distal weakness and muscle atrophy, few studies have investigated the possible key determinants of muscle quality in these patients. Therefore, the aim of this study was to evaluate circulating Irisin levels in a population of 20 CMT patients as well the association of Irisin with biochemical parameters and muscle quality. In addition, the investigators compared these data with unpublished data previously obtained in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of Charcot-Marie-Tooth disease

Exclusion Criteria:

* osteoporosis
* intestinal malabsorption
* chronic inflammatory diseases
* chronic renal failure
* severe heart failure
* neoplastic diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with Charcot-Marie-Tooth disease who have given informed consent
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-11-02 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Irisin level assessment | At enrollment
  Irisin levels in the blood at enrollment
muscle mass assessment | At enrollment
  Muscle mass determined by bioelectrical impedance analysis
muscle strenght assessment | At enrollment
  Muscle strenght by handgrip dynamometer
muscle quality assessment | At enrollment
  Muscle quality determined by bioelectrical impedance analysis
Correlation between irisin levels and muscle mass, muscle strenght, and muscle quality | Immediately after enrollment
  Correlation determined by Pearson's correlation for linear regression analysis

CONTACTS AND LOCATIONS:
Overall Officials: Michele Barone, prof., Principal Investigator — University of Bari
Locations (1):
- Policlinic Hospital, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grandis M, Shy ME. Current Therapy for Charcot-Marie-Tooth Disease. Curr Treat Options Neurol. 2005 Jan;7(1):23-31. doi: 10.1007/s11940-005-0003-5. PMID 15610704
- [Result] Mann DC, Hsu JD. Triple arthrodesis in the treatment of fixed cavovarus deformity in adolescent patients with Charcot-Marie-Tooth disease. Foot Ankle. 1992 Jan;13(1):1-6. doi: 10.1177/107110079201300101. PMID 1577335
- [Result] Guyton GP, Mann RA. The pathogenesis and surgical management of foot deformity in Charcot-Marie-Tooth disease. Foot Ankle Clin. 2000 Jun;5(2):317-26. PMID 11232233
- [Result] Corrado B, Ciardi G, Bargigli C. Rehabilitation Management of the Charcot-Marie-Tooth Syndrome: A Systematic Review of the Literature. Medicine (Baltimore). 2016 Apr;95(17):e3278. doi: 10.1097/MD.0000000000003278. PMID 27124017
- [Result] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Result] Ma J, Chen K. The role of Irisin in multiorgan protection. Mol Biol Rep. 2021 Jan;48(1):763-772. doi: 10.1007/s11033-020-06067-1. Epub 2021 Jan 3. PMID 33389537
- [Result] Maak S, Norheim F, Drevon CA, Erickson HP. Progress and Challenges in the Biology of FNDC5 and Irisin. Endocr Rev. 2021 Jul 16;42(4):436-456. doi: 10.1210/endrev/bnab003. PMID 33493316
- [Result] Colaianni G, Storlino G, Sanesi L, Colucci S, Grano M. Myokines and Osteokines in the Pathogenesis of Muscle and Bone Diseases. Curr Osteoporos Rep. 2020 Aug;18(4):401-407. doi: 10.1007/s11914-020-00600-8. PMID 32514668
- [Result] Colaianni G, Notarnicola A, Sanesi L, Brunetti G, Lippo L, Celi M, Moretti L, Pesce V, Vicenti G, Moretti B, Colucci S, Grano M. Irisin levels correlate with bone mineral density in soccer players. J Biol Regul Homeost Agents. 2017 Oct-Dec,;31(4 suppl 1):21-28. PMID 29181953
- [Result] Colaianni G, Faienza MF, Sanesi L, Brunetti G, Pignataro P, Lippo L, Bortolotti S, Storlino G, Piacente L, D'Amato G, Colucci S, Grano M. Irisin serum levels are positively correlated with bone mineral status in a population of healthy children. Pediatr Res. 2019 Mar;85(4):484-488. doi: 10.1038/s41390-019-0278-y. Epub 2019 Jan 15. PMID 30683930
- [Result] Faienza MF, Brunetti G, Sanesi L, Colaianni G, Celi M, Piacente L, D'Amato G, Schipani E, Colucci S, Grano M. High irisin levels are associated with better glycemic control and bone health in children with Type 1 diabetes. Diabetes Res Clin Pract. 2018 Jul;141:10-17. doi: 10.1016/j.diabres.2018.03.046. Epub 2018 Apr 19. PMID 29679630
- [Result] Palermo A, Sanesi L, Colaianni G, Tabacco G, Naciu AM, Cesareo R, Pedone C, Lelli D, Brunetti G, Mori G, Colucci S, Manfrini S, Napoli N, Grano M. A Novel Interplay Between Irisin and PTH: From Basic Studies to Clinical Evidence in Hyperparathyroidism. J Clin Endocrinol Metab. 2019 Aug 1;104(8):3088-3096. doi: 10.1210/jc.2018-02216. PMID 30759249
- [Result] Colaianni G, Errede M, Sanesi L, Notarnicola A, Celi M, Zerlotin R, Storlino G, Pignataro P, Oranger A, Pesce V, Tarantino U, Moretti B, Grano M. Irisin Correlates Positively With BMD in a Cohort of Older Adult Patients and Downregulates the Senescent Marker p21 in Osteoblasts. J Bone Miner Res. 2021 Feb;36(2):305-314. doi: 10.1002/jbmr.4192. Epub 2020 Oct 29. PMID 33053231
- [Result] Chang JS, Kim TH, Nguyen TT, Park KS, Kim N, Kong ID. Circulating irisin levels as a predictive biomarker for sarcopenia: A cross-sectional community-based study. Geriatr Gerontol Int. 2017 Nov;17(11):2266-2273. doi: 10.1111/ggi.13030. Epub 2017 Apr 10. PMID 28394089
- [Result] Budziareck MB, Pureza Duarte RR, Barbosa-Silva MC. Reference values and determinants for handgrip strength in healthy subjects. Clin Nutr. 2008 Jun;27(3):357-62. doi: 10.1016/j.clnu.2008.03.008. Epub 2008 May 2. PMID 18455840
- [Result] Kim HJ, So B, Choi M, Kang D, Song W. Resistance exercise training increases the expression of irisin concomitant with improvement of muscle function in aging mice and humans. Exp Gerontol. 2015 Oct;70:11-7. doi: 10.1016/j.exger.2015.07.006. Epub 2015 Jul 13. PMID 26183690
- [Derived] Colaianni G, Oranger A, Dicarlo M, Lovero R, Storlino G, Pignataro P, Fontana A, Di Serio F, Ingravallo A, Caputo G, Di Leo A, Barone M, Grano M. Irisin Serum Levels and Skeletal Muscle Assessment in a Cohort of Charcot-Marie-Tooth Patients. Front Endocrinol (Lausanne). 2022 May 12;13:886243. doi: 10.3389/fendo.2022.886243. eCollection 2022. PMID 35634506